CLINICAL TRIAL: NCT07259629
Title: Fasting Induced Hypoglycaemia in Anaesthetised Paediatric Patients
Acronym: FIGS
Status: Recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Evelina London Children's Charity (Unknown); Nova Biomedical (Industry); Kings Health Partners (Other)
Responsible Party: Sponsor
Other Study IDs: 329701
Record Dates: First submitted 2024-07-16; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Hypoglycemia; Iatrogenic; Anesthesia; Pediatrics
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fasting is a requirement to safely anesthetise patients referred for elective procedure, using the traditional 6/4/2 rule (6h for solid food or formula milk, 4h for breast milk and 2h for clear fluids), applied to all patients regardless of their age or weight. Reducing the aspiration risk however puts young children at higher risk of hypoglycemia due to the immaturity of their endocrine system and absence of metabolic reserves. The Association of Paediatric Anaesthetists of Great Britain and Ireland recommends that during day case surgery the majority of children may be given fluids without dextrose, provided blood glucose is monitored. Recent statements recommend continuing fluids until 1h before the procedure or even to give fluids when anesthetists sent for the patients. Hypoglycemia is rare in children above 2 years of age. Although the definition of hypoglycemia can differ, a threshold of 3.6mmol/l is often used given the potential neurological harm existing below this value. There is no consensus on the definition of hypoglycemia in children being fasted prior to general anesthesia, nor when nor how to treat it. Measurements are done for complex surgeries or patients deemed at risk according to the anesthetists. An audit was run in 2017 at the " Evelina London Children's Hospital ", Guy's and St Thomas' National Health Service Foundation Trust, identifying 8% of children below 2 years of age as hypoglycemic. Recent review of our Incident Reporting Systems identified 3 cases, in otherwise fit and healthy children, referred for colonoscopy with initial hypoglycemia followed by rebound hypoglycemia after management. There is an urgent need to establish a clear definition of hypoglycemia and investigate risk factors in paediatric patients referred for elective procedures under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* All American Society of Anesthesiology score (ASA) 1 - 3 children aged 1 month to 18 years presenting for an elective procedure involving general anaesthesia during the defined study period
* All elective cases, day cases will be included (patient's admitted the night before for bowel preparation prior to elective colonoscopy should also be included)
* Planned expedited cases in ASA 1 / 2 children should be included, for example nail bed repairs, lacerations, foreign body (in ear / eye / nose), simple fractures for manipulation under anesthesia / k-wires
* MRI, radiology and dental cases will be included provided the patient receives a general anaesthetic

Exclusion Criteria:

* Children aged less than 1 month
* Procedures performed under oral sedation or local anaesthesia only
* ASA status 4 and 5
* Children with any endocrine or metabolic condition or who have a fasting plan prior to general anaesthesia for glucose control:
* Type 1 or 2 diabetes mellitus, medium chain acetyl Co-enzyme A, maple syrup urine disease, glycogen storage disease, galactosaemia, urea cycle defects, familial hypercholesterolaemia, congenital disorders of glycosylation, lysosomal storage disorders, organic acidaemias, mitochondrial disorders, adrenal gland disorders, adrenoleukodystrophy, growth disorders, lipid disorders, multiple endocrine neoplasia type 1 and 2, pituitary disorders.
* Emergency and oncology procedures as these children will have different risk factors for hypoglycaemia
* Anaesthetic involvement in critically ill children e.g. airway management in emergency department, pediatric intensive care unit
* Children on glucose containing intravenous solutions or total parenteral nutrition pre-operatively
* Children on systemic steroid treatment (oral / intravenous). Children on inhalers / topical steroids should be included

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patients fasting for a procedure under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 6580 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-01-12 (Estimated)

PRIMARY OUTCOMES:
Clinical definition if hypoglycemia | Immediately/within five minutes after anesthesia induction
  Blood glucose values triggering a response from the anaesthetists with initiation of a hypoglycaemia treatment following a blood glucose measurement during anaesthetic induction

SECONDARY OUTCOMES:
4mmol/l as a suitable threshold of hypoglycemia | Immediately/within five minutes after anesthesia induction
  Number of patient with a blood glucose measurement below 4mmol/l and being treated as hypoglycaemic by an anaesthetist following a blood glucose measurement during anaesthetic induction
Distribution of glycemic measurements in fasting children | Immediately/within five minutes after anesthesia induction
  Blood glucose values in children undergoing elective procedure under general anaesthesia.
Age as a risk factor of hypoglycaemia | Immediately/within five minutes after anesthesia induction
  Number of children below 24 months of age reported as hypoglycaemic by an anaesthetist following a blood glucose measurement during anaesthetic induction
Weight as a risk factor of hypoglycaemia | Immediately/within five minutes after anesthesia induction
  Number of children weighing less than 10kg and considered as hypoglycaemic by an anaesthetist following a blood glucose measurement during anaesthetic induction
Distribution of blood ketone measurements in children fasting | Immediately/within five minutes after anesthesia induction
  Blood ketone values in children undergoing elective procedure under general anaesthesia.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter, Devon
  - Moorfields Eye Hospital, London
  - Evelina London Children's Hospital, London

IPD SHARING:
Plan to Share IPD: No